CLINICAL TRIAL: NCT04375306
Title: Resting Full-cycle Flow Ratio (RFR) Versus Angiography to Guide Revascularization Strategy in Patients Undergoing Coronary Artery By-pass Grafting (CABG): RFR-CABG Trial
Brief Title: Resting Full-cycle Flow Ratio (RFR) Versus Angiography to Guide Revascularization Strategy in Patients Undergoing Coronary Artery By-pass Grafting (CABG)
Acronym: RFR-CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9333
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
Keywords: RFR guided CABG; angiography guided CABG; Graft dysfunction
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: International prospective randomized multicenter superiority trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: All patients will undergo RFR and FFR measurement before CABG. RFR and FFR values will be blinded to the patients in both arms. In the control arm (angiography guided CABG) the RFR values will be blinded to the cardiothoracic surgeon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- angiography guided CABG (Active Comparator): angiography guided CABG
  Interventions: Procedure: Angio guided CABG
- RFR guided CABG (Experimental): RFR guided CABG
  Interventions: Procedure: RFR guided CABG

INTERVENTIONS:
Procedure: RFR guided CABG — All patients will undergo RFR and FFR measurement before CABG. RFR and FFR values will be blinded to the patients. In the experimental arm the decision to revascularize will be based on RFR.
  Arms: RFR guided CABG
Procedure: Angio guided CABG — All patients will undergo RFR and FFR measurement before CABG. RFR and FFR values will be blinded to the patients. In the control arm the RFR values will be blinded to the cardiothoracic surgeon.
  Arms: angiography guided CABG

SUMMARY:
Different trials have shown that fractional flow reserve (FFR) could successfully guide revascularization in patients undergoing percutaneous coronary intervention (PCI).

It is conceivable that a similar revascularization guidance could be useful also for surgical revascularization i.e. coronary by-pass graft (CABG). Experience learns that grafts placed on vessels with hemodynamically non-significant stenosis often occlude due to competitive antegrade flow.

Resting full-cycle Flow Ratio (RFR) is a measurement performed to evaluate the hemodynamic severity of coronary stenosis. Differently from FFR which is a measurement performed in maximal hyperemia, the RFR is a measurement that is performed in rest and therefore may predict better than FFR the baseline equilibriums that could lead to graft failure, while it has similar capacity to identify hemodynamically significant stenosis as FFR. It is unknown whether RFR guided CABG revascularization is superior as compared to angiography alone.

ELIGIBILITY:
Inclusion Criteria:

* All patients between 18 or older undergoing CABG
* Patients willing and capable to provide written informed consent

Exclusion Criteria:

* Previous CABG
* Concomitant severe valvular disease intervention
* Remaining (expected) coronary stenosis of > 50% diameter stenosis distally to graft anastomosis
* Left ventricular ejection fraction <30%
* Known transmural myocardial infarction
* Documented microvascular disease
* RFR/FFR measurement judged impossible
* Life expectancy <2 years
* Participation in other investigational clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who deceased, had a Myocardial Infarction (MI), Clinically-Driven Target Vessel Revascularization (CD-TVR), Stroke or Graft Dysfunction at 3 months post CABG | 3 months

SECONDARY OUTCOMES:
Cut-off value for the RFR that best predicts graft occlusion | Baseline
Number of participants with graft dysfunction at 3 months post CABG | 3 months
Major adverse cardiac or cerebrovascular event (MACCE), a composite of Death, MI, CD-TVR and Stroke at 1 year | 1 year
Major adverse cardiac or cerebrovascular event (MACCE), a composite of Death, MI, CD-TVR and Stroke at 3 years | 3 years
CD-TVR at 3 months post CABG | 1 year
CD-TVR at 1 year post CABG | 1 year
CD-TVR at 3 years post CABG | 3 years

CONTACTS AND LOCATIONS:
Locations (4):
- Belgium (2):
  - Imelda ziekenhuis, Bonheiden
  - AZ Sint-Jan Brugge, Bruges
- Medical University of Silesia, Katowice, Poland
- SUSCCH, Banská Bystrica, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided
This has not been decided yet.